CLINICAL TRIAL: NCT01820702
Title: Short Term Bed Rest Study: Evaluation of the Use of Artificial Gravity, Induced by Short-arm Centrifugation or the Appliance of Definite Combined Training Program to Counteract Effects of Bed Rest (Acronym: SAG Study)
Brief Title: Short Term Bed Rest Study: Evaluation of the Use of Artificial Gravity, Induced by Short-arm Centrifugation
Acronym: SAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DLR German Aerospace Center (Other)
Collaborators: European Space Agency (Other); University Hospital, Angers (Other Government); Politecnico di Milano (Other); University Hospital, Bonn (Other); University of Zurich (Other); Leiden University Medical Center (Other); German Sport University, Cologne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Contract 22126/08/NL/VJ (SAG)
Record Dates: First submitted 2012-12-11; First posted 2013-03-29 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Bone Diseases, Metabolic; Acid-Base Imbalance; Muscular Atrophy; Sprains and Strains; Protein Metabolism; Body Weight Changes; Cardiovascular Abnormalities
Keywords: bone metabolism; acid base balance; bed rest
MeSH Terms: conditions — Bone Diseases, Metabolic; Acid-Base Imbalance; Muscular Atrophy; Sprains and Strains; Body Weight Changes; Cardiovascular Abnormalities

ARMS (2):
- defined training programme (Active Comparator)
  Interventions: Other: Defined Training Programme
- Control (No Intervention)

INTERVENTIONS:
Other: Defined Training Programme — A Smith Machine with fixed rails was used to guide the heel raise and squat exercises in the vertical axis. A metronome was used to direct the subjects during the performance of the exercises. Squats and heel raises were performed against body weight plus the additional weight of the barbell (15 kg). The heel raises were performed with straight knees and without ankle dorsiflexion. The shallow squats were performed continuously for 3 minutes. The hopping and the cross-hopping exercises were performed without Smith Machine. The bilateral hops were performed at ~ 3 repetitions per second with 15-s rest insertions between each set. Cross-hopping was performed continuously for 3 minutes against ~ 1.3 repetitions per second. Except for the duration of the static squat, with progressed from 45 s at HDT1 to 70 s at HDT5, none of the exercises were progressed during the study. Including the scheduled rest pauses, the LRT sessions were completed in 24 minutes.
  Arms: defined training programme

SUMMARY:
Randomized cross-over design with 10 male subjects and 3 campaigns to test whether the negative effects of bed rest (6º head-down tilt) on the various systems of the body and the consequences to health of simulated weightlessness can be counteracted by the use of a defined training programme.

DETAILED DESCRIPTION:
The SAG study was a single center, open-label crossover trial with healthy men conducted in three campaigns at the Institute of Aerospace Medicine, Cologne, Germany.

The subjects were quasi randomized alternatively by enrolment to undertake the different training interventions or to be in the control group during 5 days of immobilisation in 6° head down tilt position. The subjects were quasi randomized either to the one of the training programs or the non-training group depending on the arrival at the Institute of Aerospace Medicine.

The study started November 01st, 2010 and was finished May 29th, 2011. The first campaign lasted from November 01st to November 21sh, 2010, the second campaign from January 10th to January 30th, 2011 and the third campaign from May 09th to May 29th, 2011.

Each campaign comprised a 5 day adaptation-, a 5 day intervention phase in HDT bed rest, and a 5 day recovery phase (15 days in total) in-house at the Metabolic Ward of the Institute of Aerospace Medicine.

Baseline Data were collected during the adaptation phase (BDC Baseline Data Collection) when subjects could move free inside the lab. The intervention was administered during the bed rest phase where the subjects had to lie in bed in 6° head down tilt (HDT Head Down Tilt) position and were not allowed to get up. Recumbency was to be adhered to at all times including all activities (hygienic procedures, leisure activities). The bed rest phase was followed by a recovery phase (R+).

ELIGIBILITY:
Inclusion Criteria:

* • Healthy male test subjects, aged between 20 and 45 years old with a Body Mass Index (BMI) of 20 - 26 kg/m2 and a height of 158 - 190 cm (62 - 75 inches)

  * 65 - 85 kg
  * Not a competitive athlete
  * Non-smoker, for at least six months before the start of the study
  * In the position to participate in the complete study
  * Demonstrable social insurance and official certificate of absence of criminal record
  * Successful completion of screening examination
  * Provision of Declaration on Consent at the start of the study

Exclusion Criteria:

* • Drug, medication or alcohol abuse (regular consumption of more than 20-30 g alcohol/day)

  * Smoking
  * Vegetarian, vegan
  * Migraine
  * Previous psychiatric illness
  * Claustrophobia
  * Hiatus hernia
  * Gastro-oesophageal reflux
  * Diabetes mellitus
  * Rheumatic illness
  * Muscle or joint disorder
  * Prolapse of intervertebral disk
  * Pronounced orthostatic intolerance
  * Hyperlipidaemia (deviations from standard values, standard values: TG < 180 mg/dl, cumulative CH < 200 mg/dl, HDL > 35 mg/dl, LDL < 160 mg/dl)
  * Renal dysfunction (deviation from plasma creatinin standard values, standard value < 1.20 mg/dl)
  * Thyroid dysfunction (deviation from standard values for plasma TSH, standard value TSH 0.27 - 4.20 U/l)
  * Hyperhomocysteinemia (deviation from standard value for plasma homocysteine, standard value homocysteine >15 µmol/l)
  * Hyper-, Hypouricemia (deviation from plasma uric acid standard values, age dependent standard value 3.0-6.9 mg/dl)
  * Hyper-, Hypocalcemia (deviation from plasma calcium standard values, age dependent standard value 2.15-2.64 mmol/l)
  * Anaemia: (< as standard values for plasma haemoglobin, standard values for men 13.5-17.5 g/dl)
  * Iron deficiency: ferritin < 30 µg/l
  * Vitamin D deficiency: D3-25-OH < 50 ng/ml
  * Blood gas values deviating from the normal values:

    * pH 7.38-7.42
    * pCO2 34-45 mmHg
    * pO2 79-98 mmHg
    * HCO3 20-28 mmol/l
    * Base deviation ± 2 mmol/l
  * Family history of thrombosis or positive response in thrombosis screening procedure: Biochemical analysis of the following parameter: ATIII, protein C and S activities, factor V Leiden, prothrombin mutants, lupus PTT
  * Chronic back complaints
  * Bone fracture in the year preceding the study
  * Bone density of the femur and lower spine (L1-L4) 1.5 SD ≤ t-score
  * Metal implants or other kinds of bone synthesis materials
  * Participation in another clinical study within the last 2 months before start of this study
  * Imprisoned at the time of the study
  * Any other condition which makes the test subject unsuitable for study inclusion in the opinion of the examiner

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Maximal knee extensor and plantar flexor muscle force | Baseline, after 5 days of bed rest
  The maximal voluntary isometric force (MVC) was assessed before and following bed rest. MVC measurements were obtained from the left leg using the Biodex 3 system (Biodex Medical Systems, Shirley, New York, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Mulder, Dr., Study Director — German Aerospace Center
Locations (1):
- German Aerospace Center (DLR), Cologne, Germany